CLINICAL TRIAL: NCT06615479
Title: A Phase 3, Randomized, Open-Label, Multicenter Study to Compare the Efficacy and Safety of Arlocabtagene Autoleucel (BMS-986393), a GPRC5D-directed CAR-T Cell Therapy, Versus Standard Regimens in Adult Participants With Relapsed or Refractory and Lenalidomide-exposed Multiple Myeloma
Brief Title: A Study to Compare the Efficacy and Safety of BMS-986393 Versus Standard Regimens in Adult Participants With Relapsed or Refractory and Lenalidomide-exposed Multiple Myeloma (QUINTESSENTIAL-2)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA088-1007
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Relapsed or Refractory Multiple Myeloma (RRMM)
Keywords: Relapsed or Refractory Multiple Myeloma; Multiple Myeloma; BMS-986393; Chimeric Antigen Receptor T-cell (CAR T-cell); CAR T-cell Therapy; Arlocabtagene Autoleucel; Arlo-cel
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Cyclophosphamide; fludarabine; daratumumab; pomalidomide; Dexamethasone; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: BMS-986393; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Daratumumab; Drug: Pomalidomide; Drug: Dexamethasone; Drug: Carfilzomib
- Arm B (Active Comparator)
  Interventions: Drug: Daratumumab; Drug: Pomalidomide; Drug: Dexamethasone; Drug: Carfilzomib

INTERVENTIONS:
Drug: BMS-986393 — Specified dose on specified days
  Other Names: Arlo-cel
  Arms: Arm A
Drug: Cyclophosphamide — Specified dose on specified days
  Arms: Arm A
Drug: Fludarabine — Specified dose on specified days
  Arms: Arm A
Drug: Daratumumab — Specified dose on specified days
Drug: Pomalidomide — Specified dose on specified days
Drug: Dexamethasone — Specified dose on specified days
Drug: Carfilzomib — Specified dose on specified days

SUMMARY:
The purpose of this study is to compare the efficacy and safety of arlo-cel (BMS-986393) versus standard regimens in adult participants with Relapsed or Refractory and Lenalidomide-exposed Multiple Myeloma.

ELIGIBILITY:
Inclusion Criteria

* Participants must have relapsed or refractory multiple myeloma (RRMM).
* Participants must have received at least 1 but no greater than 3 prior multiple myeloma (MM) regimens which may include a proteasome inhibitor (PI), an immunomodulatory drug (IMiD), and an anti-CD38 monoclonal antibody and have prior exposure to lenalidomide.
* Participants must have a documented diagnosis of MM as per International Myeloma Working Group Criteria.
* Participants must have measurable disease during screening.
* Participants must have adequate organ function.
* Participants must have an Eastern Cooperative Oncology group performance status 0 or 1.

Exclusion Criteria

* Participants must not have known active or history of central nervous system (CNS) involvement of Multiple Myeloma (MM).
* Participants must not have solitary plasmacytomas or non-secretory myeloma without other evidence of measurable disease.
* Participants must not need urgent treatment due to rapidly progressing MM.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2032-06-22 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 5 years after the last participant is randomized
Minimal residual disease (MRD)-negativity in complete response (CR) | Up to 1 year after the last participant is randomized

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years after the last participant is randomized
Overall response rate (ORR) | Up to 5 years after the last participant is randomized
Minimal residual disease (MRD)-negative status | Up to 5 years after the last participant is randomized
Complete response rate (CRR) | Up to 5 years after the last participant is randomized
Time to response (TTR) | Up to 5 years after the last participant is randomized
Duration of response (DOR) | Up to 5 years after the last participant is randomized
Maximum observed concentration (Cmax) of transgene level | Up to 5 years after the last participant is randomized
Time of maximum observed plasma concentration (Tmax) of transgene level | Up to 5 years after the last participant is randomized
Area under the concentration-time curve (AUC) of transgene level | Up to 5 years after the last participant is randomized
Changes from baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire- Core 30 items (QLQ-C30) primary domains | Up to 5 years after the last participant is randomized
  EORTC QLQ-C30 primary domains: fatigue, pain, physical functioning, role functioning, cognitive functioning, and global health status/quality of life (QoL).
Changes from baseline in EORTC Quality of Life Multiple Myeloma Module- 20 items (QLQ-MY20) primary domains | Up to 5 years after the last participant is randomized
  EORTC QLQ-MY20 primary domains: disease symptoms and side effects of treatment
Time to meaningful improvement in EORTC QLQ-C30 global health status/QoL. | Up to 5 years after the last participant is randomized

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (137):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCLA Hematology/Oncology - Santa Monica, Los Angeles, California
  - Local Institution - 0050, Orange, California
  - Local Institution - 0223, Washington D.C., District of Columbia
  - Local Institution - 0231, Jacksonville, Florida
  - Local Institution - 0130, Miami, Florida
  - Local Institution - 0228, Orlando, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Louisiana State University Health Sciences Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Local Institution - 0219, Minneapolis, Minnesota
  - Local Institution - 0229, New York, New York
  - Local Institution - 0221, Stony Brook, New York
  - Local Institution - 0067, Charlotte, North Carolina
  - Local Institution - 0216, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Local Institution - 0232, Pittsburgh, Pennsylvania
  - Local Institution - 0227, Charleston, South Carolina
  - Local Institution - 0184, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Local Institution - 0195, Milwaukee, Wisconsin
- Argentina (3):
  - Hospital Italiano de Buenos Aires, ABB, Buenos Aires F.D.
  - Local Institution - 0214, ABB, Buenos Aires F.D.
  - Hospital Aleman, Buenos Aires, Buenos Aires F.D.
- Australia (8):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Local Institution - 0190, Liverpool, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Health, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (2):
  - Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria
  - Hanusch-Krankenhaus, Vienna
- Belgium (4):
  - Antwerp University Hospital, Edegem, Antwerpen
  - Local Institution - 0217, Brussels, Bruxelles-Capitale, Région de
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant-Godinne - Site Godinne, Yvoir, Namur
  - UZ Gent, Ghent, Oost-Vlaanderen
- Brazil (4):
  - Local Institution - 0012, Nova Lima, Minas Gerais
  - Local Institution - 0013, São Paulo, São Paulo
  - Local Institution - 0103, São Paulo, São Paulo
  - Local Institution - 0031, São Paulo
- Canada (5):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - QEII Health Sciences Centre - Victoria General Site, Halifax, Nova Scotia
  - Local Institution - 0192, Hamilton, Ontario
  - CIUSSS de l'Est-de-l'Île-de-Montréal, Montreal, Quebec
- Czechia (3):
  - Fakultní nemocnice Brno Bohunice, Brno, Brno-město
  - Local Institution - 0093, Hradec Králové, Hradec Králové
  - Vseobecna fakultni nemocnice v Praze, Prague
- Denmark (4):
  - Rigshospitalet, Copenhagen, Capital Region
  - Aarhus Universitetshospital, Skejby, Aarhus, Central Jutland
  - Roskilde Sygehus, Roskilde, Region Sjælland
  - Odense Universitetshospital, Odense, Region Syddanmark
- Finland (3):
  - Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus), Helsinki, Uusimaa
  - Oulun yliopistollinen sairaala, Oulu
  - Turku University Hospital, Turku
- France (5):
  - Hopital Claude Huriez - CHU de Lille, Lille, Nord
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes, Pays de la Loire Region
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhône
  - Henri Mondor Hospital, Créteil, Val-de-Marne
  - Hôpital Saint-Louis, Paris
- Germany (11):
  - TUM Klinikum, Munich, Bavaria
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Klinikum Chemnitz - Flemmingstraße, Chemnitz, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitaetsklinikum Magdeburg, Magdeburg, Saxony-Anhalt
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel, Schleswig-Holstein
  - Charité Campus Virchow-Klinikum, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Klinikum Nuernberg Nord, Nuremberg
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (3):
  - University Hospital of Patras, Pátrai, Achaḯa
  - Evangelismos General Hospital of Athens, Athens, Attikí
  - Attikon General University Hospital, Chaïdári, Attikí
- Hungary (2):
  - Debreceni Egyetem Klinikai Kozpont, Debrecen, Hajdú-Bihar
  - Local Institution - 0125, Budapest
- Israel (3):
  - Sheba Medical Center, Ramat Gan, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Sourasky Medical Center, Tel Aviv, Tell Abīb
- Italy (6):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Turin, Piedmont
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Ospedale San Martino, Genova
  - Local Institution - 0106, Udine
- Japan (10):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Hyogo Medical University Hospital, Nishinomiya, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kyushu University Hospital, Fukuoka
  - Kumamoto University Hospital, Kumamoto
  - National Hospital Organization Okayama Medical Center, Okayama
  - Osaka Red Cross Hospital, Osaka
  - Japanese Red Cross Medical Center, Tokyo
  - Yamagata University Hospital, Yamagata
- Netherlands (4):
  - Radboudumc, Nijmegen, Gelderland
  - Maastricht UMC+, Maastricht, Limburg
  - Amsterdam UMC, locatie VUmc, Amsterdam, North Holland
  - Universitair Medisch Centrum Utrecht, Utrecht
- Sykehusapoteket Ull, Oslo, Norway
- Poland (4):
  - Centrum Onkologii Ziemi Lubelskiej, Lublin, Lublin Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Local Institution - 0084, Katowice
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz, Łódź Voivodeship
- Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto, Portugal
- Romania (2):
  - Fundeni Clinical Institute, Bucharest, București
  - Institutul Regional de Oncologie, Iași
- Local Institution - 0178, Riyadh, Saudi Arabia
- Singapore (2):
  - National University Hospital, Singapore, Central Singapore
  - Local Institution - 0181, Singapore, Central Singapore
- South Korea (4):
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (6):
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruña [La Coruña]
  - Hospital Universitari Son Espases, Palma, Balears [Baleares]
  - Institut Catalan d Oncologia (ICO) - Badalona, Badalona, Barcelona [Barcelona]
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Virgen Nieves, Granada
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
- Sweden (2):
  - Karolinska Universitetssjukhuset Huddinge, Huddinge
  - Skånes Universitetssjukhus Lund, Lund
- Switzerland (2):
  - Inselspital Bern, Bern, Canton of Bern
  - Cantonal Hospital St.Gallen, Sankt Gallen, Canton of St. Gallen
- Taiwan (4):
  - National Taiwan University Cancer Center (NTUCC), Taipei City, Taipei
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Local Institution - 0200, Taipei
- Local Institution - 0170, Ankara, Turkey (Türkiye)
- United Kingdom (5):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - University College London Hospital, London, London, City of
  - Churchill Hospital, Oxford, Oxfordshire
  - The Christie NHS Foundation Trust, Manchester
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06615479.html